CLINICAL TRIAL: NCT01007006
Title: Evaluation of a Telepharmacy Robotic Medicine Delivery Unit in Warrior Transition Unit Patients With Traumatic Brain Injury, Post-Traumatic Stress Disorder, or Polytrauma
Brief Title: Telepharmacy Robotic Medicine Delivery Unit "TRMDU" Assessment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to gain approval from commanding Army and Navy officers to conduct study.
Sponsor: University of Illinois at Chicago (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Daniel R. Touchette, Professor of Pharmacy, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009-0936; W81XWH-09-1-0092 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Traumatic Brain Injury; Posttraumatic Stress Disorders; Trauma; Combat Disorders; Pain
Keywords: Telepharmacy Robotic Medicine Delivery Unit; Brain Injuries; Stress Disorders; Combat disorders; Polytrauma; Adherence
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Wounds and Injuries; Combat Disorders; Pain; Brain Injuries; Stress Disorders, Traumatic; Multiple Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMRDU (Experimental): Telepharmacy Robotic Medicine Delivery Unit (TMRDU) group will receive TMRDU plus medication management
  Interventions: Device: TMRDU
- Control (No Intervention): Control arm will receive only medication management, no TMRDU.

INTERVENTIONS:
Device: TMRDU — The TMRDU will assist study subjects with taking their medications as prescribed by notifying them when the next dose is due and tracking whether and when it was taken.
  Other Names: Electronic Medication Management Assistant, (EMMA) (R)
  Arms: TMRDU

SUMMARY:
The objective of this study is to evaluate whether use of TRMDU in addition to medication review leads to improved outcomes and reduced health care costs for patients when compared with medication review alone. The study will be conducted in patients assigned to Department of Defense (DOD) Warrior Transition Units (WTU's), similar DOD units, and VA polytrauma centers.

DETAILED DESCRIPTION:
The military has been witnessing an increased number of patients with combat related impairments such as traumatic brain injury, post traumatic stress disorder and polytrauma which has lead to sub optimal medication self management. TRMDU is a medical device developed by INRange Systems Inc. that delivers medications and emits a sound alert to assist the patient. It can be used in a hospital, clinic, or residential setting. It can be remotely accessed by the health care professionals, and it allows physicians and other prescribers to remotely change scheduling or adjust prescriptions.

Use of TRMDU in hospital settings is expected to improve outcomes by improving medication self management, increasing adherence, reducing medication errors, and thereby associated costs. Further, it may contribute to overall improvement in a patient's psychological well-being and quality of life.

ELIGIBILITY:
Inclusion Criteria: Subjects must be

* At least 18 years of age
* Alert and oriented to person , place and time
* Primarily use English language for written and oral communication
* Have diagnosis of Traumatic Brain Injury(TBI) Multiple Traumatic Brain Injury (MTBI), Post Traumatic Stress Disorder (PTSD) or Polytrauma.
* Taking at least 4 chronic prescription medications
* Living in a participating WTU or enrolled in Tampa Veterans Administration polytrauma outpatient treatment facility at the time of enrollment
* Achieve a minimum score of 24 on Mini-Mental State Examination

Exclusion Criteria: If patients meet following criteria they are excluded from the study

* Disabilities preventing safe use of the TRMDU
* Projected life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12 (Estimated); Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Adherence | Six months
  Pill counts and self report (Morisky 8-item)

SECONDARY OUTCOMES:
Intensity and type of pain | Three months
  Short-Form McGill Pain Questionnaire; 15 descriptors rated on intensity of 0=none to 3=severe
Psychological well-being | Three months
  Profile of Moods Brief Scale; scores of 6 subscales range from 0-20, with higher scores indicating higher distress, except for one subscale which is negatively scored.
Health related quality of life | Three months
  Short-Form 36; 8 domains of general health with higher scores indicating less disability
Total cost of care | Six months
  Six-month medication and medical cost of care will be extracted from the DOD prescription and medical claims databases

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Touchette, MA, Principal Investigator — University of Illinois at Chicago; Jill M Winters, PhD, Principal Investigator — Columbia College of Nursing
Locations (3):
- United States (3):
  - Naval Hospital Camp Pendleton, Camp Pendleton, California
  - James A Haley VA Hospital and Polytrauma Facility, Tampa, Florida
  - Ireland Army Community Hospital, Fort Knox, Kentucky

REFERENCES:
- [Background] Bates DW. Preventing medication errors: a summary. Am J Health Syst Pharm. 2007 Jul 15;64(14 Suppl 9):S3-9; quiz S24-6. doi: 10.2146/ajhp070190. PMID 17617512
- [Background] Cantor JB, Ashman T, Gordon W, Ginsberg A, Engmann C, Egan M, Spielman L, Dijkers M, Flanagan S. Fatigue after traumatic brain injury and its impact on participation and quality of life. J Head Trauma Rehabil. 2008 Jan-Feb;23(1):41-51. doi: 10.1097/01.HTR.0000308720.70288.af. PMID 18219234
- [Background] Ernst FR, Grizzle AJ. Drug-related morbidity and mortality: updating the cost-of-illness model. J Am Pharm Assoc (Wash). 2001 Mar-Apr;41(2):192-9. doi: 10.1016/s1086-5802(16)31229-3. PMID 11297331
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Background] Institute for Healthcare Improvement. (2009). Prevent adverse drug events (medication reconciliation).
- [Background] Krousel-Wood M, Islam T, Webber LS, Re RN, Morisky DE, Muntner P. New medication adherence scale versus pharmacy fill rates in seniors with hypertension. Am J Manag Care. 2009 Jan;15(1):59-66. PMID 19146365
- [Background] Lee JK, Grace KA, Taylor AJ. Effect of a pharmacy care program on medication adherence and persistence, blood pressure, and low-density lipoprotein cholesterol: a randomized controlled trial. JAMA. 2006 Dec 6;296(21):2563-71. doi: 10.1001/jama.296.21.joc60162. Epub 2006 Nov 13. PMID 17101639
- [Background] McDonald HP, Garg AX, Haynes RB. Interventions to enhance patient adherence to medication prescriptions: scientific review. JAMA. 2002 Dec 11;288(22):2868-79. doi: 10.1001/jama.288.22.2868. PMID 12472329
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Nathan A, Goodyer L, Lovejoy A, Rashid A. 'Brown bag' medication reviews as a means of optimizing patients' use of medication and of identifying potential clinical problems. Fam Pract. 1999 Jun;16(3):278-82. doi: 10.1093/fampra/16.3.278. PMID 10439982
- [Background] O'Connor PJ. Improving medication adherence: challenges for physicians, payers, and policy makers. Arch Intern Med. 2006 Sep 25;166(17):1802-4. doi: 10.1001/archinte.166.17.1802. No abstract available. PMID 17000934
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Sakthong P, Chabunthom R, Charoenvisuthiwongs R. Psychometric properties of the Thai version of the 8-item Morisky Medication Adherence Scale in patients with type 2 diabetes. Ann Pharmacother. 2009 May;43(5):950-7. doi: 10.1345/aph.1L453. Epub 2009 Apr 14. PMID 19366872
- [Background] Svarstad BL, Chewning BA, Sleath BL, Claesson C. The Brief Medication Questionnaire: a tool for screening patient adherence and barriers to adherence. Patient Educ Couns. 1999 Jun;37(2):113-24. doi: 10.1016/s0738-3991(98)00107-4. PMID 14528539
- [Background] Touchette DR, Burns AL, Bough MA, Blackburn JC. Survey of medication therapy management programs under Medicare part D. J Am Pharm Assoc (2003). 2006 Nov-Dec;46(6):683-91. doi: 10.1331/1544-3191.46.6.683.touchette. PMID 17176683
- [Background] van Mil JW, Westerlund LO, Hersberger KE, Schaefer MA. Drug-related problem classification systems. Ann Pharmacother. 2004 May;38(5):859-67. doi: 10.1345/aph.1D182. Epub 2004 Mar 30. PMID 15054145
- [Background] Vasterling JJ, Proctor SP, Amoroso P, Kane R, Heeren T, White RF. Neuropsychological outcomes of army personnel following deployment to the Iraq war. JAMA. 2006 Aug 2;296(5):519-29. doi: 10.1001/jama.296.5.519. PMID 16882958
- [Background] Institute for Healthcare Improvement. (2009).
- [Background] Burkhart PV, Sabate E. Adherence to long-term therapies: evidence for action. J Nurs Scholarsh. 2003;35(3):207. No abstract available. PMID 14562485
- [Background] McNair, D., M. Lorr, et al. (1992). POMS Manual
- [Background] National Council on Patient Information and Education. (2008).
- [Background] Ware, J. E., K. K. Snow, et al. (1993). SF36 health survey: Manual and interpretation guide. Boston. MA, New England Medical Center
- See also: National Council on Patient Information and Education. (2008). "Public policy & adherence." Retrieved July 20, 2008 — http://www.talkaboutrx.org/documents/enhancing_prescription_medicine_adherence.pdf